CLINICAL TRIAL: NCT01452191
Title: Keeping Children Safe at Home: Cluster Randomised Controlled Trial of the Implementation of an Injury Prevention Briefing in Children's Centres for the Prevention of Fire-related Injuries
Brief Title: Helping Children's Centres to Enhance Home Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11007
Record Dates: First submitted 2011-10-10; First posted 2011-10-14 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-05

CONDITIONS: Burns; Smoke Inhalation Injury
Keywords: Cluster Randomised Controlled Trial; Community Health Services; prevention & control; Accidents, Home; Child Health Services
MeSH Terms: conditions — Burns; Smoke Inhalation Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Injury Prevention Briefing and facilitation (Active Comparator): Children's Centres will be given an Injury Prevention Briefing which offers guidance on best evidence on reducing fire related injuries in the home, and facilitation by the research team to support implementation of the IPB
  Interventions: Behavioral: Injury Prevention Briefing Plus facilitation
- Injury Prevention Briefing only (Active Comparator): Children's Centres will be given an Injury Prevention Briefing (IPB) , which offers guidance on best evidence on reducing fire related injuries in the home.
  Interventions: Behavioral: Injury Prevention Briefing
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Injury Prevention Briefing Plus facilitation — Injury Prevention Briefing (IPB) to provide best evidence on what works to reduce house fire injuries, and activities to get the evidence into practice. This arm will receive facilitation to support the implementation of the information in the IPB
  Arms: Injury Prevention Briefing and facilitation
Behavioral: Injury Prevention Briefing — Children's centres will receive the Injury Prevention Briefing only.
  Arms: Injury Prevention Briefing only

SUMMARY:
Many children have accidents, some are very serious and they are a major cause of death in children aged 1-4 years. Many accidents are preventable This study aims to find out the best way to help Children's Centres to provide home safety information about preventing fires to parents and carers of young children.

36 Children's Centres in four study centres, Nottingham, Bristol, Norwich and Newcastle will be recruited to the study. 30 families will be recruited from each Children's Centre. Children's Centres serving the most deprived populations will be eligible to take part.

Families will be eligible to take part if they have attended a participating Children's Centre in the previous three months, have parents who are 16 years or older, have a child under three years old and live within the catchment area of that Children's Centre. When 30 families have been recruited that Centre will be allocated, at random, to one of three groups. Children's Centres in group one will be provided with guidance about preventing fire-related injuries (an Injury Prevention Briefing (IPB))and help and support to implement the IPB, the second group will be sent the IPB and the third group will not be provided with the IPB ('usual care'). Children's Centres will devise their own programmes of safety advice for parents based on the IPB.

At recruitment and 12 months later, families and Children's Centres will complete questionnaires about fire safety practices. Children's Centres will also complete a paper-based tool about the implementation process at 12 months. Information about barriers and facilitators to implementing the IPB will be collected through interviews with Children's Centre staff.

The study will run from May 2011 to March 2014.

ELIGIBILITY:
Inclusion Criteria:

There are two levels of participation, Children's Centres as participants, who will be delivering the intervention, and families as participants, who will be receiving the intervention.

Children's Centres:

Phase 1 Children's Centres in the four study areas (Nottingham, Newcastle, Bristol and Norwich) Phase 2 Children's Centres in more disadvantaged areas (defined as those who have more than 50% of under 5 year-old children in their Centre catchment area who live in one of the 30% most disadvantaged Super Output Areas).

Families Any family who has attended the participating Children's Centre in the previous three months, who have a child under three years old, and lives within the catchment area of that Children's Centres.

Exclusion Criteria:

Children's Centres:

Phase 2 Children's Centres that are not in more disadvantaged areas as defined above and phase 3 or subsequent wave Children's Centres.

Families Families who attend a participating Children's Centre who do not have any children under the age of 3 years Any parent who is under-16 years of age.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1112 (Actual)
Dates: Start 2011-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Kendrick, Principal Investigator — University of Nottingham
Locations (4):
- United Kingdom (4):
  - University of West of England, Bristol, Bristol
  - Newcastle University, Newcastle
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - University of Nottingham, Nottingham

REFERENCES:
- [Derived] Ploubidis GB, Edwards P, Kendrick D; Keeping Children Safe Study Group. Measuring behaviours for escaping from house fires: use of latent variable models to summarise multiple behaviours. BMC Res Notes. 2015 Dec 15;8:789. doi: 10.1186/s13104-015-1769-5. PMID 26670153
- [Derived] Hindmarch P, Hawkins A, McColl E, Hayes M, Majsak-Newman G, Ablewhite J, Deave T, Kendrick D; Keeping Children Safe study group. Recruitment and retention strategies and the examination of attrition bias in a randomised controlled trial in children's centres serving families in disadvantaged areas of England. Trials. 2015 Mar 7;16:79. doi: 10.1186/s13063-015-0578-4. PMID 25886131
- [Derived] Deave T, Towner E, McColl E, Reading R, Sutton A, Coupland C, Cooper N, Stewart J, Hayes M, Pitchforth E, Watson M, Kendrick D. Multicentre cluster randomised controlled trial evaluating implementation of a fire prevention Injury Prevention Briefing in children's centres: study protocol. BMC Public Health. 2014 Jan 22;14:69. doi: 10.1186/1471-2458-14-69. PMID 24450931

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Children's centres
Groups:
- Injury Prevention Briefing and Facilitation: Children's Centres will be given an Injury Prevention Briefing which offers guidance on best evidence on reducing fire related injuries in the home, a three hour staff training session and facilitation by the research team to support implementation of the IPB.
- Injury Prevention Briefing Only: An Injury Prevention Briefing (IPB) , which offers guidance on best evidence on reducing fire related injuries in the home, will be posted to Children's centres.
- Usual Care: Children's centres undertake usual fire prevention activity.
Period: Overall Study
Arm/Group | Injury Prevention Briefing and Facilitation | Injury Prevention Briefing Only | Usual Care
Started | 373; 12 Children's centres | 369; 12 Children's centres | 370; 12 Children's centres
Completed | 241; 12 Children's centres | 252; 12 Children's centres | 258; 12 Children's centres
Not Completed | 132; 0 Children's centres | 117; 0 Children's centres | 112; 0 Children's centres

BASELINE CHARACTERISTICS:
Population: Families nested within Children's centres
Units Other Than Participants: Children's centres
Groups:
- Total: Total of all reporting groups
Arm/Group | Injury Prevention Briefing and Facilitation | Injury Prevention Briefing Only | Usual Care | Total
Number analyzed (Participants) | 373 | 369 | 370 | 1112
Number analyzed (Children's centres) | 12 | 12 | 12 | 36
Age, Customized [Count of Participants; unit: Participants] — Maternal age, dichotomised as 20 years and younger or over 20 years Population: Number differs from overall number where baseline data was missing
  Participants
    number analyzed (Participants) | 356 | 350 | 354 | 1060
    Maternal age 20 years or younger | 20 | 17 | 17 | 54
Sex/Gender, Customized [Number; unit: participants] — Sex was not measured in the trial Population: Sex was not measured in the trial
  participants
    number analyzed (Participants) | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Family ethnicity reported as White British Population: Number differs from overall number where baseline data is missing
  Participants
    number analyzed (Participants) | 361 | 351 | 350 | 1062
    Family ethnicity White Bristish: Ethnicity: White British | 348 | 323 | 337 | 1008
    Family ethnicity White Bristish: Ethnicity: Other ethnic group | 13 | 28 | 13 | 54
Region of Enrollment [Number; unit: participants]
  United Kingdom | 373 | 369 | 370 | 1112
Family have a plan for escaping from a house fire [Count of Participants; unit: Participants] — Population: Number differs fromoverall number where baseline data is missing
  Participants
    number analyzed (Participants) | 366 | 364 | 363 | 1093
    (all) | 149 | 153 | 159 | 461
Lead agency for Children's centre [Count of Units; unit: Children's centres]
  Local Authority | 9 | 7 | 10 | 26
  NHS | 2 | 0 | 0 | 2
  Voluntary sector | 1 | 5 | 2 | 8
Ofsted score for overall effectiveness of Children's centre [Count of Units; unit: Children's centres] — Population: Number differs from overall number where baseline data is missing
  Children's centres
    number analyzed (Children's centres) | 11 | 12 | 12 | 35
    Outstanding | 4 | 2 | 3 | 9
    Good/satisfactory | 7 | 10 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Families With a Fire Escape Plan (Ascertained From Self-completion Questionnaire).
Time Frame: 1 year
Population: Data on this outcome was missing for 5 participants in the Injury Prevention Briefing and Facilitation arm, 9 in the Injury Prevention Briefing only arm and 4 in the Usual Care arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Injury Prevention Briefing and Facilitation | Injury Prevention Briefing Only | Usual Care
Number analyzed (Participants) | 236 | 243 | 254
Participants | 120 | 108 | 119

2. Secondary Outcome: The Number of Childrens Centres Providing Information and Advice on Smoke Alarms
Time Frame: 1 year
Population: Analysis based at level of Children's centres. Data on this outcome was missing for one Children's centre in the Injury Prevention Briefing only arm.
Measure: Count of Units; unit: Children's centres
Units Other Than Participants: Children's centres
Arm/Group | Injury Prevention Briefing and Facilitation | Injury Prevention Briefing Only | Usual Care
Number analyzed (Participants) | 241 | 252 | 258
Number analyzed (Children's centres) | 12 | 11 | 12
Children's centres | 11 | 11 | 11

3. Secondary Outcome: The Number of Children's Centres Providing Information and Advice on How to Make a Fire Escape Plan
Time Frame: 1 year
Population: Analysis at level of Children's centres. Data on this outcome was missing for one Children's centre in the Usual Care arm.
Measure: Count of Units; unit: Children's centres
Units Other Than Participants: Children's centres
Arm/Group | Injury Prevention Briefing and Facilitation | Injury Prevention Briefing Only | Usual Care
Number analyzed (Participants) | 241 | 252 | 258
Number analyzed (Children's centres) | 12 | 12 | 11
Children's centres | 12 | 9 | 8

4. Secondary Outcome: The Number of Children's Centres Providing Information and Advice on the Causes of House Fires
Time Frame: 1 year
Population: Analysis at level of Children's centres
Measure: Count of Units; unit: Children's centres
Units Other Than Participants: Children's centres
Arm/Group | Injury Prevention Briefing and Facilitation | Injury Prevention Briefing Only | Usual Care
Number analyzed (Participants) | 241 | 252 | 258
Number analyzed (Children's centres) | 12 | 12 | 12
Children's centres | 12 | 12 | 11

5. Secondary Outcome: The Number of Children's Centres Providing Information and Advice on Child Behaviour and Fire Prevention
Time Frame: 1 year
Measure: Count of Units; unit: Children's centres
Units Other Than Participants: Children's centres
Arm/Group | Injury Prevention Briefing and Facilitation | Injury Prevention Briefing Only | Usual Care
Number analyzed (Participants) | 241 | 252 | 258
Number analyzed (Children's centres) | 12 | 12 | 12
Children's centres | 12 | 11 | 8

6. Secondary Outcome: The Number of Children's Centres Providing Information and Advice on Bedtime Routines to Prevent Fires
Time Frame: 1 year
Population: Analysis at level of Children's centres. Data on this outcome was missing for one Children's centre in the Injury Prevention Briefing and Facilitation arm and one Children's centre in the Usual Care arm.
Measure: Count of Units; unit: Children's centres
Units Other Than Participants: Children's centres
Arm/Group | Injury Prevention Briefing and Facilitation | Injury Prevention Briefing Only | Usual Care
Number analyzed (Participants) | 241 | 252 | 258
Number analyzed (Children's centres) | 11 | 12 | 11
Children's centres | 11 | 8 | 5

ADVERSE EVENTS:
Arm/Group | Injury Prevention Briefing and Facilitation | Injury Prevention Briefing Only | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/373 | 0/369 | 0/370
Other Adverse Events (participants affected / at risk) | 0/373 | 0/369 | 0/370

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No